CLINICAL TRIAL: NCT03265496
Title: Correlation Between Tissue and Plasmatic EGFR in CBNPC With EGFR Mutation or Predictive Factor of EGFR Mutation
Acronym: CONCORDE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of recruted patient was not sufficient
Sponsor: Centre Oscar Lambret (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CONCORDE-1510
Record Dates: First submitted 2017-08-14; First posted 2017-08-29 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Nsclc
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Liquid Biopsy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study procedure (Experimental): Clinical exam. Liquid biopsy. Diagnostic exam (biopsy and imagery). 1st line treatment. tumor evaluation. Biopsy
  Interventions: Procedure: Clinical exam; Procedure: Liquid biopsy; Procedure: Diagnostic exam; Drug: 1st line treatment; Procedure: tumor evaluation; Biological: Biopsy

INTERVENTIONS:
Procedure: Clinical exam — Clinical exam is performed before treatment start
Procedure: Liquid biopsy — Liquid biopsy will be performed at baseline and every 3 cycles of chemotherapy until progression disease
Procedure: Diagnostic exam — Diagnostic exam (biopsy and imagery exam) will be performed at baseline if not previously done or incompletely done.
Drug: 1st line treatment — 1st line chemotherapy (chemotherapy or EGFR targeted therapy) will be performed until progression disease.
  Other Names: 1st line chemotherapy
Procedure: tumor evaluation — Tumor evaluation will be performed every 3 cycles of chemotherapy
Biological: Biopsy — Biopsy will be performed at the end of study, after progression disease, if a mutation of EGFR is detected in tumor DNA.

SUMMARY:
Condorde main objective is to evaluate the correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed on ctDNA after liquid biopsy. EGFR status will be assessed by real time PCR (rtPCR), digital PCR (dPCR) and Next Generation Sequencing (NGS) in patients with chemotherapy naive lung carcinoma.

DETAILED DESCRIPTION:
Newest therapeutic breakthrough are often based on molecular analysis of tumoral tissue before treatment initiation or after emergence of resistance. Tumoral tissue is commonly obtained by biopsy. However, tumor biopsy is an invasive, scarcely repeatable and costly technics. Moreover, tumor samples, obtained by biopsy, doesn't represent tumor heterogeneity and cannot inform about tumor evolution over time.

Recent improvement have been done in detection and characterization of blood circulating tumoral DNA (ctDNA). ctDNA reach regularly the blood stream after tumoral cell apoptosis or necrosis and could be extract and sequenced by some molecular biology technics such as real time PCR (rtPCR), digital PCR (dPCR) or next generation sequencing (NGS). Interesting, Several studies demonstrate that some genomic alterations of solid cancer can be characterized after sequencing of ctDNA. Other experiments pointed that ctDNA level could be linked to tumor stage and patient prognostic.

These progress lead to the development of a new non invasive method for extraction of ctDNA called liquid biopsy (LB). LB could be useful for monitor tumoral genotype, assess tumor response to treatment and detect residual tumor cells after curative treatment. Moreover LB could be an essential method for study of tumor cells molecular alterations mechanisms during targeted cancer therapies, when clinical resistance occurs.

Non-small cell lung cancer (NSCLC) is the most frequently diagnosticated type of lung cancer. Regular first line chemotherapy is based on the use of platinum salts. However, some mutations in the EGFR gene could add sensitivity of NSCLC to tyrosine kinase inhibitors such as gefitinib, erlotinib or afatinib. Consequently, the search for molecular mutations in genome of NSCLC cells is of prior interest for patients with clinically advanced NSCLC.

Recently, some studies demonstrate that mutational EGFR status of NSCLC was sharply correlated between tumoral tissue, obtained by classical biopsy, and ctDNA, collected by liquid biopsy.

These results provide promising data encouraging the use of LB for study of NSCLC ctDNA. However some experimentations are needed to ensure these data.

For that reason, CONCORDE clinical trial will evaluate the correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy. EGFR status will be assessed by real time PCR (rtPCR), digital PCR (dPCR) and Next Generation Sequencing (NGS) in patients with chemotherapy naive lung carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years
* Metastatic lung carcinoma
* With: - EGFR gene mutation
* Or at least 2 predictive factors of addictive mutation (Women, non smocking or cessation > 3 years, Asiatic, lung adenocarcinoma)
* Eligible for 1st line treatment
* Performance status ≤ 3
* Available tumor sample or tumor reachable for biopsy
* With informed and signed consent
* Affiliation to the National Social Security System

Exclusion Criteria:

* Previous radiotherapy treatment in months preceding initials samples
* Pregnant or breastfeeding women
* Patient not able to give consent or unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy. At diagnostic. NGS. | Baseline
  For patient with mutant EGFR. Evaluate, by next generation sequencing at diagnostic, the correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy.

SECONDARY OUTCOMES:
Correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy. At diagnostic. rtPCR. | Baseline
  For patient with mutant EGFR. Evaluate, by real time PCR at diagnostic, the correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy.
Correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy. At diagnostic. dPCR. | Baseline
  For patient with mutant EGFR. Evaluate, by digital PCR at diagnostic, the correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy.
Correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy. At disease progression. NGS. | From Baseline to disease progression, up to 2 years
  For patient with mutant EGFR. Evaluate, by Next Generation Sequencing at disease progression, the correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy.
Correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy. At disease progression. rtPCR. | From Baseline to disease progression, up to 2 years
  For patient with mutant EGFR. Evaluate, by rtPCR at disease progression, the correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy.
Correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy. At disease progression. dPCR. | From Baseline to disease progression, up to 2 years
  For patient with mutant EGFR. Evaluate, by dPCR at disease progression, the correlation between EGFR mutational status determined after tumor biopsy and EGFR mutational status analyzed after liquid biopsy.
Incidence of oncogenic mutation for patients with predictive factors | From Baseline to disease progression, up to 2 years
  To evaluate the incidence of oncogenic mutations in populations with clinical predictive factors of these mutations.
Predictive value of ctDNA during treatment with EGFR targeting therapy. | From Baseline to disease progression, up to 2 years
  To assess the predictive value of mutant ctDNA during treatment with EGFR targeting therapy.
Mutations on ctDNA and tumor biopsy. | From Baseline to disease progression, up to 2 years
  To search for mutations leading to treatment resistance on ctDNA and tumor biopsy at proved disease progression

OTHER OUTCOMES:
Mutation in ctDNA | From Baseline to disease progression, up to 2 years
  To detect, at early stage, mutations on liquid biopsy. To identify, at early stage, mutations leading to treatment resistance by Next Generation Sequencing.
expression pattern of tumor grade and resistance | From Baseline to disease progression, up to 2 years
  To identify a predictive expression pattern for grade and treatment resistance of tumor by iterative sampling during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kotecki Nuria, MD, Principal Investigator — Centre Oscar Lambret; Cortot Alexis, Pr, Principal Investigator — CHRU LILLE
Locations (2):
- France (2):
  - Centre Oscar Lambret, Lille
  - CHRU Lille, Lille

IPD SHARING:
Plan to Share IPD: No